CLINICAL TRIAL: NCT04670575
Title: Vivity Outcomes in Patients With Early Stage Glaucoma
Acronym: VIVA
Status: Completed | Type: Observational
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Other Study IDs: VIVA
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma; Cataract; Presbyopia
Keywords: Extended Range of Vision, Intraocular Lens Technology, Glaucoma
MeSH Terms: conditions — Glaucoma; Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vivity: Patients implanted with Vivity or Vivity Toric intraocular lens at the time of cataract surgery.
  Interventions: Procedure: Cataract Surgery with Implantation of Vivity Extended Range of Vision IOL

INTERVENTIONS:
Procedure: Cataract Surgery with Implantation of Vivity Extended Range of Vision IOL — Patients with early stage glaucoma implanted with Vivity or Vivity Toric IOL

SUMMARY:
The goal of the study is to determine the visual outcomes in patients with mild, pre-perimetric glaucoma who undergo cataract surgery with implantation of the Alcon Vivity Extended Range Intraocular Lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least age 45 years of age undergoing uncomplicated cataract surgery with optional concomitant minimally invasive glaucoma surgery (MIGS)
2. Subjects with documented diagnosis of pre-perimetric glaucoma
3. Calculated lens power within Vivity/Vivity toric range
4. Willing and able to comprehend informed consent and complete 4-6 month post-op visit
5. Potential postoperative BCDVA of 20/20 or better in each eye based on Investigator's medical opinion

Exclusion Criteria:

1. Ocular comorbidity, other than pre-perimetric glaucoma, that could reduce the potential postoperative BCDVA
2. Previous ocular surgery including refractive surgery
3. Subjects who are pregnant or plan to become pregnant during the course of the study.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with early stage glaucoma with cataracts in both eyes who are planned to have bilateral cataract surgery with implantation of Vivity or Vivity Toric intraocular lens.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity | 4-6 months
Uncorrected Intermediate Visual Acuity | 4-6 months
Uncorrected Near Visual Acuity | 4-6 months

SECONDARY OUTCOMES:
Contrast Sensitivity | 4-6 months
  As measured by Pelli Robson Chart
Patient Satisfaction and Spectacle Independence Survey Results | 4-6 months
Mean Refractive Spherical Equivalent | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Shafer, MD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No